CLINICAL TRIAL: NCT06835023
Title: A Randomized Controlled Trial Evaluating Fluid Resuscitation in Acute Pancreatitis: Dextran 40 and Ringer's Lactate (1:3 Ratio) Versus Ringer's Lactate Alone
Brief Title: Dextran 40 Plus Ringer's Lactate Vs. Ringer's Lactate Alone for Fluid Resuscitation in Acute Pancreatitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Satu Mare County Emergency Hospital (Other Government)
Responsible Party: Principal Investigator, COSTEA CRISTIAN, PHD STUDENT DOCTOR, Satu Mare County Emergency Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE15/14.10.2021; 27/11.10.2021 (Other: Ethics Committee of Satu Mare County Hospital)
Record Dates: First submitted 2025-02-01; First posted 2025-02-19 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Acute Pancreatitis (AP); Acute Pancreatic Fluid Collection; Fluid Resuscitation
Keywords: Fluid resuscitation; Acute pancreatitis; Dextran; Ringer Lactat solution; combination colloid-crystalloid
MeSH Terms: conditions — Pancreatitis | interventions — Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dextran 40 plus Ringer Lactat 1:3 ratio (Experimental): 50 patients with acute pancreatitis will receive Dextran 40 plus RInger Lactat 1:3 ratio early to admission in the hospital
  Interventions: Drug: Dextran+Ringer Lactat(D+RLS)
- Ringer Lactat (Active Comparator): 50 patients will receive only Ringer Lactat
  Interventions: Drug: Ringer lactate (RLS)

INTERVENTIONS:
Drug: Ringer lactate (RLS) — 50 patients will receive only Ringer Lactat
  Arms: Ringer Lactat
Drug: Dextran+Ringer Lactat(D+RLS) — 50 patients Dextran+RInger Lactat 1:3 ratio
  Arms: Dextran 40 plus Ringer Lactat 1:3 ratio

SUMMARY:
This clinical trial aims to learn if a combination of Dextran 40 and Ringer's lactate solution can improve fluid resuscitation in mild and moderate acute pancreatitis (AP) and prevent complications. The main questions it aims to answer are:

Does early fluid resuscitation with Dextran 40 plus Ringer's lactate improve patient outcomes compared to Ringer's alone? Does this treatment reduce inflammation, organ failure, and the need for intensive care unit (ICU) admission? Researchers will compare Dextran 40 plus Ringer's lactate to Ringer's alone to see if the combination therapy is more effective in reducing disease severity and complications.

Participants will:

Receive either Dextran 40 plus Ringer's lactate (1:3 ratio) or Ringer's lactate alone.

Have blood tests every 24 hours to measure inflammation and organ function. Be monitored for changes in disease severity, need for ICU admission, and hospitalization duration.

This study will help determine the best fluid resuscitation strategy for treating mild and moderate acute pancreatitis.

DETAILED DESCRIPTION:
Detailed Description Acute pancreatitis (AP) is a common gastrointestinal disorder requiring hospitalization, with an incidence of approximately 40 cases per 100,000 individuals. The severity of AP ranges from mild to severe, with 15-20% of cases progressing to severe acute pancreatitis (SAP), which is characterized by organ failure and local complications. The mortality rate for severe acute pancreatitis remains high, reaching 20-30%, highlighting the critical need for early and adequate fluid resuscitation in emergency settings.

Despite universal recommendations for early-volume resuscitation, there is no clear consensus regarding the optimal fluid type, infusion rate, total volume, or monitoring strategy. Fluid resuscitation's primary objective is to prevent or minimize systemic inflammatory response syndrome (SIRS), which significantly contributes to AP progression.

This randomized controlled trial (RCT) will compare the effectiveness of a colloid-crystalloid combination (Dextran 40 in sodium chloride [NaCl] 0.9 grams per liter [g/L] solution and Ringer's lactate solution in a 1:3 ratio) versus Ringer's lactate solution alone in preventing disease progression and reducing complications in patients with mild or moderate AP.

Study Design This randomized clinical trial (RCT) will be conducted at Satu Mare County Emergency Hospital and enroll approximately 100 patients diagnosed with mild or moderate AP.

Fluid Administration Rate: 1,5 mL/kg/h, based on patient hemodynamic status.

* Data Collection and Assessment
* Clinical and Demographic Data:
* Age, sex.
* Lifestyle factors (alcohol consumption, smoking).
* Symptom onset time and severity classification (based on the Revised Atlanta -Classification, 2012).

  =Diagnostic Criteria (Requires ≥2 of 3):
* Acute upper abdominal pain.
* Serum amylase/lipase levels ≥3 times the upper standard limit (ULN).
* Imaging findings (CT, ultrasound, or MRI) consistent with AP.

Organ Failure Assessment:

-Modified Marshall Scoring System (2012).

Severity Scoring:

* Modified Glasgow Score.
* Acute Physiology and Chronic Health Evaluation II (APACHE II).
* Bedside Index for Severity in Acute Pancreatitis (BISAP).
* CT Severity Index.

Laboratory Biomarkers & Monitoring

Blood samples will be collected at admission and every 24 hours to assess:

* Pancreatic Enzymes: Amylase, lipase.
* Inflammatory Markers & Organ Function Parameters:
* C-reactive protein (CRP).
* Erythrocyte sedimentation rate (ESR).
* Hematocrit.
* Urea, creatinine.
* Systemic inflammatory response syndrome (SIRS) markers.
* Fibrinogen, ferritin.
* Procalcitonin at enrollment and 72 hours.

Additional Monitoring:

An ultrasound will measure the Inferior vena cava (IVC) diameter and collapsibility index to estimate central venous pressure (CVP) and hemodynamic status.

Urine output every 24 hours (target ≥0.5 mL/kg/h as an adequate resuscitation marker).

Primary and Secondary Outcome Measures

Primary Outcomes:

Reduction in C-reactive protein (CRP) and SIRS

Secondary Outcomes:

* Reduced duration of hospitalization and lower ICU admission rates.
* Reduction of erythrocyte sedimentation rate (ESR) and other inflammatory markers.
* Complication rates (e.g., pancreatic necrosis, organ failure).
* Hospitalization costs.
* In-hospital mortality and follow-up mortality at 3 months.

Follow-up and Study Endpoints Patients will be monitored throughout hospitalization and followed up at 12 weeks post-discharge.

Expected Impact This study aims to identify the optimal fluid resuscitation strategy for mild and moderate AP. If the colloid-crystalloid combination proves superior, it could lead to changes in clinical guidelines for AP management, potentially reducing organ failure, ICU admissions, and mortality rates.

ELIGIBILITY:
Inclusion Criteria:

* adults (≥18 years) diagnosed with mild or moderate acute pancreatitis
* must provide written informed consent for study participation.

Exclusion Criteria:

* patients who decline to provide informed consent.
* patients are non-compliant with treatment and follow-up visits.
* pregnant individuals.
* patients requiring concomitant treatment that is contraindicated within the study protocol.
* patients who develop conditions that contraindicate the administration of the investigational medication.
* patients experiencing severe adverse reactions necessitating treatment discontinuation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2025-05-12 (Estimated); Study Completion 2025-05-12 (Estimated)

PRIMARY OUTCOMES:
roportion of Participants with Resolution of Systemic Inflammatory Response Syndrome (SIRS) | From enrollment (Day 1) to Day 4 or discharge, whichever occurs first.
  The percentage of participants who experience resolution of SIRS, defined as meeting ≤1 of the SIRS criteria (body temperature, heart rate, respiratory rate, and white blood cell count) for two consecutive 24-hour assessments.
  SIRS Criteria:
  * Body temperature <36°C or >38°C
  * Heart rate >90 beats per minute
  * Respiratory rate >20 breaths per minute or PaCO₂ <32 mmHg
  * White blood cell count <4,000 cells/mm³ or >12,000 cells/mm³
  Data Collection & Aggregation:
  * SIRS criteria will be assessed every 24 hours.
  * The percentage of participants achieving SIRS resolution by Day 4 or discharge will be reported.
  Unit of Measure: Percentage of participants achieving SIRS resolution.
Mean Percentage Reduction in Serum C-Reactive Protein (CRP) Levels (mg/L) from Baseline | Baseline (Day 1) to Day 4 or discharge, whichever occurs first
  Serum C-Reactive Protein (CRP) will be measured in milligrams per liter (mg/L) at baseline (Day 1) and then every 24 hours until Day 4 or discharge.
  The outcome will be calculated as the mean percentage reduction in CRP from baseline to the final recorded value.
  CRP measurements will be performed using standardized high-sensitivity assays
  Unit of Measure: Mean percentage reduction in CRP levels (mg/L).

CONTACTS AND LOCATIONS:
Locations (1):
- Spitalul Judetean de Urgenta Satu Mare, Satu Mare, Satu Mare County, Romania

IPD SHARING:
Plan to Share IPD: Yes
Patients will be randomized into two groups:
  Experimental group:
  Dextran 40 in hypertonic saline + Ringer's lactate (1:3 ratio), in addition to standard treatment.
  Control group:
  Ringer's lactate alone, in addition to standard treatment. Fluids will be administered at a controlled hydration rate (5-10 mL/kg/h).
Supporting Information: CSR
Time Frame: 12 May 2025, until 12 May 2026